CLINICAL TRIAL: NCT07050394
Title: A Dose-expansion Trial Exploring the Safety and Efficacy of Intravenous HNF4α srRNA in Patients With Unresectable Locally Advanced or Metastatic Colorectal Cancer
Brief Title: A Dose-Expansion Trial of Intravenous HNF4α srRNA for Unresectable or Metastatic Colorectal Cancer
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai Changzheng Hospital (Other)
Responsible Party: Principal Investigator, Wei-Fen Xie, Professor, Shanghai Changzheng Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CZXH-CRC-2025-IIT
Record Dates: First submitted 2025-06-17; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Colorectal Cancer Metastatic; Colorectal Cancer Recurrent; Colorectal Cancer Stage IV
Keywords: Colorectal Cancer; Hepatocyte nuclear factor 4α; Differentiation therapy
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD-GA-102 (Experimental): A lipid nanoparticle-encapsulated self-replicating RNA encoding hepatocyte nuclear factor 4α
  Interventions: Drug: CD-GA-102

INTERVENTIONS:
Drug: CD-GA-102 — CD-GA-102 will be administered intravenously at 50 μg per dose, with dosing scheduled at 2 weeks (±3 days) and 4 weeks (±3 days) after the initial dose, followed by maintenance therapy every 3 weeks (±3 days). Dosing intervals may be adjusted based on participant tolerability and safety. After receiving at least two doses of CD-GA-102 monotherapy and completing safety assessments, participants may be offered combination therapies, as determined by the investigator.

SUMMARY:
This study is a single-arm, open-label, exploratory clinical trial. Building on the previous dose-escalation trial, this dose-expansion trial aims to evaluate the safety and tolerability of intravenous monotherapy with CD-GA-102 or its combination with immunotherapy and other systemic treatments in patients with unresectable locally advanced or metastatic colorectal cancer, and to preliminarily explore its efficacy in treating colorectal cancer.

DETAILED DESCRIPTION:
In this study, CD-GA-102 will be administered via peripheral intravenous injection for the treatment of colorectal cancer at a dose of 50 μg per administration. The second dose will be given 2 weeks (±3 days) after the initial administration, and the third dose will be given 4 weeks (±3 days) after the initial administration. Subsequently, maintenance therapy will be administered every 3 weeks (±3 days). The dosing interval may be adjusted based on the participants' tolerability, safety, and therapeutic response. After receiving at least two doses of intravenous monotherapy with CD-GA-102 and completing the safety assessment following the last dose, participants may be offered combination therapy with immune checkpoint inhibitors, targeted therapy, or other systemic treatments, as determined by the investigator after a comprehensive evaluation.

Up to approximately 20 participants will be enrolled in this dose-expansion phase. Based on the results of this phase, the safety and tolerability of intravenous monotherapy with CD-GA-102 or its combination with immunotherapy and other systemic treatments will be further assessed. The antitumor activity will be evaluated according to the RECIST v1.1 criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years, regardless of gender.
2. Patients with colorectal cancer confirmed by histology or cytology.
3. Patients with unresectable locally advanced or metastatic colorectal cancer.
4. Patients who are not suitable for or intolerant of standard systemic therapy; or patients who have progressed after receiving standard systemic therapy (including but not limited to the following regimens) as confirmed by RECIST v1.1: chemotherapy based on fluorouracil, oxaliplatin, or irinotecan, and targeted drugs such as anti-VEGF/EGFR monoclonal antibodies.
5. According to RECIST v1.1, patients must have at least one measurable lesion. Lesions that have received local treatment (including surgery, radiotherapy, TACE, and ablation) cannot be selected as target lesions, unless the lesion is the only measurable lesion and has clearly progressed according to imaging, in which case it may be considered as a target lesion.
6. Life expectancy ≥ 12 weeks.
7. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) score of 0-2.
8. Fertile male participants and women of childbearing age must agree to use effective contraception from the time of signing the informed consent form until 6 months after the last dose of the investigational drug. Women of childbearing age include premenopausal women and women within 2 years of menopause. Women of childbearing age must have a negative serum pregnancy test within ≤7 days before the first dose of the investigational drug.
9. Willing to sign the written informed consent form and voluntarily comply with the protocol.

Exclusion Criteria:

1. Patients who have completed standard adjuvant chemotherapy after tumor resection and relapsed or developed metastasis after a drug-free interval of 6 months, and have not received standard systemic therapy.
2. Patients with tumor tissue testing confirming mismatch repair deficiency or high microsatellite instability (dMMR/MSI-H) who have not received immune checkpoint inhibitor treatment (PD-1 monoclonal antibody or PD-L1 monoclonal antibody).
3. Patients with clinical or radiological evidence of current intestinal obstruction, perforation, or bleeding; or patients assessed by the investigator to be at high risk of perforation or bleeding.
4. Serum albumin < 28 g/L, or bilirubin > 3×ULN, or aspartate aminotransferase (AST), alkaline phosphatase (ALP), or alanine aminotransferase (ALT) > 5×ULN.
5. Patients with significant renal impairment, serum creatinine > 1.5×ULN, or creatinine clearance < 40 mL/min; urine protein <2+ (if urine protein ≥2+, a 24-hour urine protein quantification is required, and patients with 24-hour urine protein quantification <1 g may be eligible).
6. Absolute neutrophil count < 1.5×10^9/L, or platelets < 50×10^9/L, or hemoglobin < 9 g/dL.
7. International Normalized Ratio (INR) > 2.
8. Patients with known brain metastases from tumors.
9. Patients with uncontrolled hypertension, diabetes, or other severe cardiac or pulmonary diseases, or severe organ dysfunction.
10. Patients who have received local or systemic anti-tumor treatments (including immunotherapy, targeted therapy, or chemotherapy) within 4 weeks, or radiotherapy within 3 weeks, except for treatment regimens assessed as disease progression according to RECIST (version 1.1) criteria.
11. Patients with adverse events related to previous local or systemic anti-tumor treatments still ≥ Grade 2 (excluding alopecia and other events deemed tolerable by the investigator).
12. Patients with uncontrollable active infections (e.g., pulmonary or abdominal infections).
13. Patients with malignancies other than colorectal cancer within the past 5 years, with the exception of low-risk malignancies with a low risk of metastasis or death (estimated 5-year overall survival > 90%), such as early gastrointestinal cancer treated effectively, cervical carcinoma in situ, non-melanoma skin cancer, localized prostate cancer, etc.
14. Patients with active autoimmune diseases requiring systemic therapy within the past 2 years, or autoimmune diseases judged by the investigator to have a potential for recurrence or planned treatment, including but not limited to inflammatory bowel disease, celiac disease, Wegener's granulomatosis, Hashimoto's thyroiditis, systemic lupus erythematosus, scleroderma, sarcoidosis, or autoimmune hepatitis.
15. Patients who require systemic treatment with corticosteroids (prednisone or equivalent > 10 mg/day) or other immunosuppressive drugs within 14 days before the first dose of the investigational drug.
16. Patients who are preparing for or have previously undergone allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.
17. Patients who are positive for HBV-DNA or HCV RNA.
18. Patients with known active tuberculosis. Patients suspected of having active tuberculosis must be excluded based on chest imaging, sputum tests, and clinical symptoms and signs.
19. Patients who are positive for human immunodeficiency virus (HIV).
20. Pregnant or breastfeeding women, or women who cannot rule out the possibility of pregnancy.
21. Patients who have participated in other drug trials within the past 4 weeks.
22. Other situations deemed by the investigator as unsuitable for participation in this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-06-10 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate，ORR | From the first study dose date until the date of documented complete response or partial response, assessed up to 24 months
  Evaluate the objective response rate of HNF4α srRNA monotherapy or in combination with immunotherapy and other systemic treatments in patients with metastatic colorectal cancer, according to the RECIST v1.1 criteria

SECONDARY OUTCOMES:
Safty and tolerability | Through study completion, an average of 2 years
  Evaluate the incidence and severity of adverse events (AEs), serious adverse events (SAEs), and AEs leading to treatment discontinuation associated with intravenous monotherapy of CD-GA-102 or its combination with immunotherapy and other systemic treatments
Duration of Response (DOR) | up to 24 months
  Duration of Response (DOR) evaluated according to RECIST v1.1 criteria
Progression-Free Survival，PFS | up to 24 months
  Progression-Free Survival of patients evaluated according to RECIST v1.1 criteria
Time To Progression，TTP | up to 24 months
  Time To Progression of patients evaluated according to RECIST v1.1 criteria
Time To Response，TTR | up to 24 months
  Time To Response of patients evaluated according to RECIST v1.1 criteria
Disease Control Rate，DCR | up to 24 months
  Disease Control Rate evaluated according to RECIST v1.1 criteria
Clinical Benefit Rate，CBR | up to 24 months
  Clinical Benefit Rate evaluated according to RECIST v1.1 criteria
Overall Survival，OS | Throughout the entire course of treatment until the end of the follow-up period, an average of 2 years
  Overall Survival of patients
Patient Reported Outcome-1，PRO-1 | Through study completion, an average of 2 years
  The European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire Core 30 (QLQ-C30)
Patient Reported Outcome-2，PRO-2 | Through study completion, an average of 2 years
  Functional Assessment of Cancer Therapy Colorectal Cancer (FACT-C)
Patient Reported Outcome-3，PRO-3 | Through study completion, an average of 2 years
  The Generic EuroQol Five Dimension Five Level (EQ-5D-5L) Questionnaire
Changes in tumor markers | Through study completion, an average of 2 years
  Changes in tumor markers such as Carcinoembryonic Antigen (CEA) and Carbohydrate Antigen 199 (CA199) after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Weifen Xie, MD. PhD, Principal Investigator — Naval Medical University
Locations (1):
- Shanghai Changzheng Hospital, Shanghai, None Selected, China

IPD SHARING:
Plan to Share IPD: No